CLINICAL TRIAL: NCT01265290
Title: Optimizing Diagnostics And Therapy Of Arrhythmia And Syncope Events Using Intelligent Telemetric Solutions. Diagnostics Of Syncope In Children.
Brief Title: Optimizing Diagnostics Of Syncope Events Using Intelligent Telemetric Solutions.
Acronym: TELEMARC3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Prof. Lukasz Szumowski MD PhD, Institute of Cardiology, Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UDAPOIG.01.03.01-00-068/09-00C
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: Cardiac Arrhythmia; Cardiogenic Syncope
Keywords: Cardiac arrhythmia; Cardiogenic syncope; Pediatrics; Children
MeSH Terms: conditions — Arrhythmias, Cardiac; Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemetric ECG monitoring (Experimental): Telemetric Full Disclosure ECG monitoring
  Interventions: Device: Telemetric ECG monitoring
- 24 hours standard Holter monitoring (Experimental)
  Interventions: Device: repeated 24 hours ECG Holter monitoring

INTERVENTIONS:
Device: repeated 24 hours ECG Holter monitoring — repeated 24 hours ECG Holter monitoring
  Arms: 24 hours standard Holter monitoring
Device: Telemetric ECG monitoring — Telemetric ECG full disclosure monitoring with GSM technology
  Arms: Telemetric ECG monitoring

SUMMARY:
The purpose of this study is to assess efficacy of prolonged Full Disclosure electrocardiogram (ECG) monitoring and signal analysis using advanced telemetric technology to diagnose syncope in comparison with standard diagnostic procedure

DETAILED DESCRIPTION:
Syncope can be caused by many conditions, often benign but in some cases syncope can be a symptom of severe arrhythmia. Early diagnosis of the underlying disease is very important to identify patients with severe cardiac arrhythmia to commence adequate treatment. Standard diagnostic methods such as 24 hours Holter electrocardiogram (ECG) monitoring or Event Holter do not guarantee early diagnosis of the arrhythmia. Prolonged heart rhythm recording and analysis using an automatic full disclosure telemetric device can increase probability of arrhythmia diagnosis and early administration of adequate treatment. Study patients will be diagnosed using standard Holter ECG monitoring, Event Holter or 30 days telemetric ECG monitoring. Efficacy of telemetric monitoring in diagnosis of cardiac arrhythmia will be assessed in comparison with the standard Holter monitoring and Event Holter.

ELIGIBILITY:
Inclusion Criteria:

* History of syncope
* Ability to operate the telemetric device at home
* Exclusion of underlying neurological disease
* informed consent undersigned by the parents
* informed consent undersigned by the child if over 16 years of age

Exclusion Criteria:

* Syncope with known underlying disease
* Inability to operate the telemetric device at home
* Complete Heart block
* QT>500ms
* Implantation of ICD
* Inability to comply with the study protocol

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 640 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Recording of symptomatic or life threatening arrhythmia event | within 30 days since the start of monitoring
  ECG monitoring is conducted until occurrence of symptomatic arrhythmia or life threatening arrhythmia but not longer than 30 days. Patients in the control group will have standard ECG Holter monitoring repeated twice

SECONDARY OUTCOMES:
Occurrence of silent (asymptomatic) arrhythmia event | within 30 days since the start of monitoring
1. Verification of patient self assessment based on the Quality of Life questionnaire and EHRA scale against evidence of cardiac arrhythmia occurrence | within 30 days since the start of monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szumowski, Prof. MD PhD, Study Chair — National Institute of Cardiology, Warsaw, Poland; Katarzyna Bieganowska, Prof. MD PhD, Principal Investigator — Children's Memorial Health Institute
Locations (2):
- Poland (2):
  - Medical University of Warsaw Department of Pediatric Cardiology and General Pediatrics, Warsaw
  - The Children's Memmorial Health Institute, Warsaw